CLINICAL TRIAL: NCT05257837
Title: A Gun Safety Video Can Reduce Children's Unsafe Behavior Around Real Guns: A Randomized Clinical Trial
Brief Title: Follow-up Gun Study: Can Safety Videos Mitigate Interest in Guns in Children?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Brad Bushman, Professor of Communication and Psychology, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2021B0318
Record Dates: First submitted 2021-09-20; First posted 2022-02-25 (Actual); Results first posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-10

CONDITIONS: Psychology, Social; Adolescent Behavior
Keywords: adolescent; gun; violence; media
MeSH Terms: conditions — Adolescent Behavior | interventions — Crisis Intervention

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to watch a safety video about guns or a safety video about seatbelts.
  Participants are then randomly assigned to watch a movie containing guns, or a movie not containing guns.
  Outlier data will be excluded in analysis.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants did not know which condition they were in. Participants' parents were aware of the deception (hidden gun) and what condition their children were in (gun safety or seatbelt safety; movie with or without guns). Research personnel knew conditions as well. Research assistants who transcribed recorded laboratory sessions did not know what condition they were coding (eg. what type of movie participants watched)
  Research assistants coding the recorded observational data will be blind to the conditions of the participants they are coding, as well as the experimental hypotheses of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Gun safety vid x Movie clip - guns present (Experimental): Participants in this condition will view a gun safety video featuring The Ohio State University Chief of Police about a week before coming into the lab. In the lab, they will watch a ~20 minute clip of either The Rocketeer or National Treasure featuring guns.
  Interventions: Behavioral: Gun handling behavior; Other: Debriefing
- Gun safety vid x Movie clip - guns absent (Active Comparator): Participants in this condition will view a gun safety video featuring The Ohio State University Chief of Police about a week before coming into the lab. In the lab, they will watch a ~20 minute clip of either The Rocketeer or National Treasure with the guns edited out.
  Interventions: Behavioral: Gun handling behavior; Other: Debriefing
- Seatbelt safety video x Movie clip - guns present (Active Comparator): Participants in this condition will view a seatbelt safety video about a week before coming into the lab. In the lab, they will watch a ~20 minute clip of either The Rocketeer or National Treasure featuring guns.
  Interventions: Behavioral: Gun handling behavior; Other: Debriefing
- Seatbelt safety video x Movie clip - guns absent (Active Comparator): Participants in this condition will view a seatbelt safety video about a week before coming into the lab. In the lab, they will watch a ~20 minute clip of either The Rocketeer or National Treasure featuring guns.
  Interventions: Behavioral: Gun handling behavior; Other: Debriefing

INTERVENTIONS:
Behavioral: Gun handling behavior — Children will play in an observed room for 20 minutes. Aside from a selection of toys, two real handguns will be placed in a drawer. The handguns have been modified so they cannot fire. Inside the magazine, the handgun contains no bullets. Instead, it contains a sensor that counts the number of times the trigger is pulled with sufficient force to discharge the gun. This allows us to distinguish reliably the children who pull the trigger from those who handle the gun but do not pull the trigger
Other: Debriefing — Children and their parents will be debriefed on the actual purpose of the study, including the role of the safety video and how the movie clips were edited.

SUMMARY:
The investigators' previous research has shown that children exposed to media characters with guns in movies and video games are more likely to use real guns themselves (e.g., touch them, hold them, pull the trigger). This research tests whether exposure to a gun safety video a week before the study can help counteract dangerous behavior around guns.

DETAILED DESCRIPTION:
Guns are prominent in movies that target children. An analysis of top selling films found that the depiction of guns in violent scenes in PG-13 films that target youth has increased from the level of G and PG files in 1985 when the rating was introduced, to the level of R films by 2005, to exceed the level of R films since 2012, a trend that has continued.

Research in the investigator's lab has shown that children are more likely to use guns (e.g., handle them, pull the trigger) after exposure to movie characters who use guns. The investigators replicated this study using video games, and also found that children who had taken a gun safety course were less likely to engage in dangerous behavior around firearms. However, it is difficult to draw causal inferences about the gun safety course because children were not randomly assigned to take or not take a gun safety course.

The present research will aim to reduce dangerous behavior around firearms by first exposing participants to a gun safety video recorded by The Ohio State University Chief of Police. The control video is about car safety. Children will see the videos about a week before they come into the lab.

In the lab, children will be tested in pairs. They will first watch a film clip from one of two different PG rated films, either in its original form (with guns) or with the guns edited out. After exposure to the film, participants will be placed in a room with toys, including two real unloaded guns that have been modified for safety and include a trigger pull counter.

The study uses 2 (gun safety video vs. car safety video) X 2 (movie with guns vs. movie without guns) between-subjects factorial design.

The investigators predict that children will be less likely to engage in dangerous behavior around real firearms after viewing the gun safety video than those who viewed the car safety video, even if they see a movie with guns in the lab.

ELIGIBILITY:
Inclusion Criteria:

* Age 8-12 yrs
* No prior participation in the study
* Able to schedule participation with a known peer (8-12yo).

Exclusion Criteria:

* Younger than 8 yrs old
* Older than 12 yrs old
* Prior study participation
* Could not schedule participation with a known peer (8-12yo)

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 245 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2022-10-16 (Actual); Study Completion 2022-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brad J Bushman, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared upon request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After the manuscript is accepted for publication. No expiration date.
Access Criteria: Data will be open and available to all who want to examine them.
URL: https://osf.io/b9e84/

REFERENCES:
- [Derived] Kjaervik SL, Bushman BJ. Effect of a Gun Safety Video on Children's Behavior Around Real Guns: A Randomized Clinical Trial. JAMA Pediatr. 2023 Sep 1;177(9):903-910. doi: 10.1001/jamapediatrics.2023.2397. PMID 37459089

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited via Facebook ads, ResearchMatch, and referrals by parents/guardians.
Pre-assignment Details: Of the 245 children assessed for eligibility, 19 were excluded: 13 did not arrive at the lab; 2 filled out forms incorrectly; 2 had a defective recording; 2 did not respond to follow-up.
  An additional 10 participants were excluded from final analyses due to not finding the guns in the laboratory.
  216 participants were included in the final analyses.
Period: Overall Study
Arm/Group | Gun Safety Vid x Movie Clip - Guns Present | Gun Safety Vid x Movie Clip - Guns Absent | Seatbelt Safety Video x Movie Clip - Guns Present | Seatbelt Safety Video x Movie Clip - Guns Absent
Started | 58 | 60 | 58 | 50
Completed | 54 | 58 | 54 | 50
Not Completed | 4 | 2 | 4 | 0
Not completed — Excluded (did not find the guns) | 4 | 2 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Seatbelt Safety Video x Movie Clip - Guns Absent | Seatbelt Safety Video x Movie Clip - Guns Present | Gun Safety Vid x Movie Clip - Guns Absent | Gun Safety Vid x Movie Clip - Guns Present | Total
Number analyzed (Participants) | 50 | 54 | 58 | 54 | 216
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.0 (1.4) | 10.5 (1.3) | 10.1 (1.4) | 9.4 (1.2) | 9.98 (1.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 29 | 25 | 29 | 103
  Male | 30 | 25 | 33 | 25 | 113
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 1 | 2 | 6
  Not Hispanic or Latino | 48 | 53 | 57 | 52 | 210
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 2 | 2 | 2 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 19 | 8 | 20 | 49
  White | 37 | 28 | 34 | 27 | 126
  More than one race | 7 | 4 | 12 | 5 | 28
  Unknown or Not Reported | 2 | 1 | 1 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 50 | 54 | 58 | 54 | 216
Trait Aggressiveness [Mean (Standard Deviation); unit: units on a scale] — Scale taken from: Björkqvist, K., Österman, K., & Kaukiainen, A. (1992). The development of direct and indirect aggressive strategies in males and females. In K. Björkqvist & P. Niemelä (Eds.), Of mice and women: Aspects of female aggression (pp. 51-64). Academic Press. https://doi.org/10.1016/B978-0-12-102590-8.50010-6
  Responses: 1 - rarely; 2 - sometimes; 3 - often
  8 items, score range: 8-24
  Higher score: higher aggression
  units on a scale | .55 (.5) | .36 (.3) | .49 (.4) | .45 (.4) | .46 (.4)
Gun ownership [Count of Participants; unit: Participants] — Participants' parents/guardians were asked if they had a gun in the home.
  Participants
    Firearm present in the home | 5 | 23 | 15 | 27 | 70
    No firearm present in the home | 45 | 31 | 42 | 27 | 145
    No response | 0 | 0 | 1 | 0 | 1
Estimated interest in guns [Mean (Standard Deviation); unit: units on a scale] — Prior to coming to the lab, parents/guardians provided demographic information and estimated their child's interest in guns (0=not at all interested to 4=very interested)
  units on a scale | 1.86 (1.2) | 1.52 (1.3) | 1.69 (1.3) | 1.67 (1.4) | 1.68 (1.3)
Age-appropriate movies [Mean (Standard Deviation); unit: units on a scale] — Favorite Media Questionnaire Dillon KP, Bushman BJ. Effects of exposure to gun violence in movies on children's interest in real guns. JAMA Pediatr. 2017;171(11):1057-1062
  Children gave their three favorite films and frequency of watching. Films were coded by MPAA ratings, then sorted into age-appropriate or age-inappropriate. The two measures were multiplied and averaged.
  Frequency: 1 - rarely, 2 - sometimes, 3 - often. Rating: 0 - Age appropriate (G or PG), 1 - Age inappropriate (PG13+). Scale range: 0 - 3, higher values mean more consumption of age inappropriate media.
  units on a scale | 0.85 (0.9) | 1.15 (0.9) | 1.01 (0.9) | 0.59 (0.9) | 0.90 (0.93)

OUTCOME MEASURES:

1. Primary Outcome: Behavioral: Gun Location
Description: Trained research assistants, blind to video game condition and experimental hypotheses, will independently code the play session videos. Coders will identify whether the participants found the handguns, how long the participants held the handgun, and whether or not they pulled the trigger.
Time Frame: 20 minutes play session
Measure: Count of Participants; unit: Participants
Arm/Group | Seatbelt Safety Video x Movie Clip - Guns Absent | Seatbelt Safety Video x Movie Clip - Guns Present | Gun Safety Vid x Movie Clip - Guns Absent | Gun Safety Vid x Movie Clip - Guns Present
Number analyzed (Participants) | 50 | 58 | 60 | 58
Participants
  Found guns | 50 | 54 | 58 | 54
  Didn't find guns (excluded from final analyses) | 0 | 4 | 2 | 4

2. Primary Outcome: Behavioral: Gun Location Response - Told Adult
Description: If the participants found the handguns, the coders will identify whether the participants told an adult.
Time Frame: 20 minutes play session
Measure: Count of Participants; unit: Participants
Groups:
- Seatbelt Safety Video x Movie Clip - Guns Absent: Participants in this condition watched a seatbelt safety video prior to the laboratory portion of the study. No guns in the movie clip.
- Seatbelt Safety Video x Movie Clip - Guns Present; Gun Safety Vid x Movie Clip - Guns Present: Participants in this condition watched a gun safety video prior to the laboratory portion of the study. Guns present in the movie clip.
- Gun Safety Vid x Movie Clip - Guns Absent: Participants in this condition watched a gun safety video prior to the laboratory portion of the study. No guns in the movie clip.
Arm/Group | Seatbelt Safety Video x Movie Clip - Guns Absent | Seatbelt Safety Video x Movie Clip - Guns Present | Gun Safety Vid x Movie Clip - Guns Absent | Gun Safety Vid x Movie Clip - Guns Present
Number analyzed (Participants) | 50 | 54 | 58 | 54
Participants | 6 | 5 | 18 | 20
Statistical Analysis 1: Comparison: Seatbelt Safety Video x Movie Clip - Guns Absent vs Seatbelt Safety Video x Movie Clip - Guns Present; Test type: Superiority; p < .001, t-test, 2 sided

3. Primary Outcome: Behavioral: Gun Location Response - Touched Gun
Description: If the participants found the handguns, the coders will identify whether the participants touched the handgun.
Time Frame: 20 minute play session
Measure: Count of Participants; unit: Participants
Groups:
- Seatbelt Safety Video x Movie Clip - Guns Present; Gun Safety Vid x Movie Clip - Guns Present: Participants in this condition watched a seatbelt safety video prior to the laboratory portion of the study. Guns present in the movie clip.
- Gun Safety Vid x Movie Clip - Guns Absent: Participants in this condition watched a seatbelt safety video prior to the laboratory portion of the study. No guns in the movie clip.
Arm/Group | Seatbelt Safety Video x Movie Clip - Guns Absent | Seatbelt Safety Video x Movie Clip - Guns Present | Gun Safety Vid x Movie Clip - Guns Absent | Gun Safety Vid x Movie Clip - Guns Present
Number analyzed (Participants) | 50 | 54 | 58 | 54
Participants | 37 | 33 | 26 | 18
Statistical Analysis 1: Comparison: Seatbelt Safety Video x Movie Clip - Guns Absent vs Seatbelt Safety Video x Movie Clip - Guns Present; Test type: Superiority; p < .001, t-test, 2 sided

4. Primary Outcome: Behavioral: Gun Holding Time
Description: If participants handle the gun, coders will record how long the gun was held.
Time Frame: 20 minutes play session
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Seatbelt Safety Video x Movie Clip - Guns Absent | Seatbelt Safety Video x Movie Clip - Guns Present | Gun Safety Vid x Movie Clip - Guns Absent | Gun Safety Vid x Movie Clip - Guns Present
Number analyzed (Participants) | 50 | 54 | 58 | 54
seconds | 101.42 (219.91) | 100.40 (174.47) | 53.43 (143.13) | 31.55 (95.01)
Statistical Analysis 1: Comparison: Seatbelt Safety Video x Movie Clip - Guns Absent vs Seatbelt Safety Video x Movie Clip - Guns Present; Test type: Superiority; p = .012, t-test, 2 sided

5. Primary Outcome: Behavioral: Trigger Pulled
Description: When the gun was handled, this measures whether or not the participant(s) pulled the trigger.
Time Frame: 20 minute play session
Measure: Count of Participants; unit: Participants
Arm/Group | Seatbelt Safety Video x Movie Clip - Guns Absent | Seatbelt Safety Video x Movie Clip - Guns Present | Gun Safety Vid x Movie Clip - Guns Absent | Gun Safety Vid x Movie Clip - Guns Present
Number analyzed (Participants) | 50 | 54 | 58 | 54
Participants | 17 | 14 | 7 | 3

6. Primary Outcome: Number of Trigger Pulls
Description: The two guns hidden in the playroom contain sensors that count how often the trigger is pulled with sufficient force to discharge the gun. A counter on the weapon displays the number of pulls, which will be entered into a data file along with the observational data described below. Observational data will also be used to confirm trigger pull counts.
  Note: This measure includes all 216 participants who found the handguns.
Time Frame: 20 minutes play session
Measure: Mean (Standard Deviation); unit: Trigger pulls
Arm/Group | Seatbelt Safety Video x Movie Clip - Guns Absent | Seatbelt Safety Video x Movie Clip - Guns Present | Gun Safety Vid x Movie Clip - Guns Absent | Gun Safety Vid x Movie Clip - Guns Present
Number analyzed (Participants) | 50 | 54 | 58 | 54
Trigger pulls | 7.26 (14.66) | 7.90 (17.36) | 6.41 (26.51) | 1.96 (9.55)
Statistical Analysis 1: Comparison: Seatbelt Safety Video x Movie Clip - Guns Absent vs Seatbelt Safety Video x Movie Clip - Guns Present; Test type: Superiority; p = .217, t-test, 2 sided

7. Primary Outcome: Gun Pointing With Trigger Pull
Description: Trained research assistants, blind to video game condition and experimental hypotheses, will independently code the play session videos. If participants pulled the trigger, were they pointing the gun at themselves or their partners?
  Calculations done using all participants who found a firearm.
Time Frame: 20 minute play session
Measure: Mean (Standard Deviation); unit: Trigger pulls
Arm/Group | Seatbelt Safety Video x Movie Clip - Guns Absent | Seatbelt Safety Video x Movie Clip - Guns Present | Gun Safety Vid x Movie Clip - Guns Absent | Gun Safety Vid x Movie Clip - Guns Present
Number analyzed (Participants) | 50 | 54 | 58 | 54
Trigger pulls | 2.60 (12.96) | 1.74 (8.64) | 2.34 (5.78) | 1.38 (4.83)
Statistical Analysis 1: Comparison: Seatbelt Safety Video x Movie Clip - Guns Absent vs Seatbelt Safety Video x Movie Clip - Guns Present; Test type: Superiority; p = .745, t-test, 2 sided

8. Secondary Outcome: Attitudes Toward Guns
Description: Participants will complete a post-test questionnaire that collects data on the child's attitudes towards guns. Questionnaire is a 15-item attitudes towards guns survey (e.g., "I don't like being around people with guns because someone could end up getting hurt"; 0=strongly disagree to 4=strongly agree
Time Frame: After 20 minutes play session, 5 minute questionnaire
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Seatbelt Safety Video x Movie Clip - Guns Absent | Seatbelt Safety Video x Movie Clip - Guns Present | Gun Safety Vid x Movie Clip - Guns Absent | Gun Safety Vid x Movie Clip - Guns Present
Number analyzed (Participants) | 50 | 54 | 58 | 54
units on a scale | 2.99 (0.6) | 2.82 (0.6) | 3.06 (0.6) | 3.15 (0.6)

ADVERSE EVENTS:
Time Frame: Each participant was called two weeks after the date of the study and given a follow-up survey.
Arm/Group | Seatbelt Safety Video x Movie Clip - Guns Absent | Seatbelt Safety Video x Movie Clip - Guns Present | Gun Safety Vid x Movie Clip - Guns Absent | Gun Safety Vid x Movie Clip - Guns Present
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/58 | 0/60 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/58 | 0/60 | 0/58
Other Adverse Events (participants affected / at risk) | 0/50 | 0/58 | 0/60 | 0/58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2022-01-14): https://cdn.clinicaltrials.gov/large-docs/37/NCT05257837/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2023-04-05): https://cdn.clinicaltrials.gov/large-docs/37/NCT05257837/SAP_001.pdf